CLINICAL TRIAL: NCT04162678
Title: Establishing a Diagnosis of Lung Cancer Through a Fluid Biopsy
Brief Title: Fluid Biopsy for the Diagnosis of Lung Cancer
Status: Terminated | Type: Observational
Why Stopped: insufficient accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2N-19-3; NCI-2019-05861 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2N-19-3 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diagnostic (blood collection via fluid biopsy, lab analysis): Patients undergo collection of blood samples on day 1 for analysis via HD-SCA fluid biopsy. Medical charts of patients are reviewed at 3 months post-biopsy or CT screening.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Procedure: Liquid Biopsy; Other: Medical Chart Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood via HD-SCA fluid biopsy
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Liquid Biopsy — Undergo collection of blood via HD-SCA fluid biopsy
  Other Names: Plasma Biopsy
Other: Medical Chart Review — Review of medical chart
  Other Names: Chart Review

SUMMARY:
This trial collects and studies blood samples via fluid biopsy for the diagnosis of lung cancer. Studying blood samples in the laboratory may help doctors develop a blood test for lung cancer in the future and provide a better way to screen patients for lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the sensitivity and specificity of the fluid biopsy in establishing a diagnosis of bronchogenic carcinoma.

SECONDARY OBJECTIVES:

I. To determine the accuracy of determination of the histologic subtype of bronchogenic lung cancer.

II. To determine the relative contribution of cell based high definition circulating tumor cell assay (HD-CTC) and imaging mass cytometry (IMC) and plasma based circulating tumor deoxyribonucleic acid (ctDNA) assays in determination of diagnosis and histologic subtype.

OUTLINE:

Patients undergo collection of blood samples on day 1 for analysis via high definition (HD)-single cell analysis (SCA) fluid biopsy. Medical charts of patients are reviewed at 3 months post-biopsy or computed tomography (CT) screening.

After completion of study, patients are followed for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo a diagnostic biopsy for possible lung cancer or
* Completed a diagnostic lung cancer biopsy in the prior 2 weeks and has not yet undergone treatment or
* Planning or completed in the last 2 weeks a CT lung cancer screen
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study
* Known other solid tumor malignancy other than lung cancer requiring ongoing active treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a biopsy or CT screening for lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Clinical diagnosis of lung cancer | Within 90 days of tissue biopsy
  Descriptive statistics including sensitivity, specificity, positive, and negative predictive value will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge J Nieva, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California